CLINICAL TRIAL: NCT01110096
Title: Randomised Controlled Clinical Trial Comparing Two Family Interventions to Treat Obesity in Children Between 7 and 12 Years.
Brief Title: Family Based Intervention in Childhood obesitY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: St. Olavs Hospital (Other); Røros Rehabiliteringssenter (Unknown); Oslo University Hospital (Other); Evjeklinikken (Other); Gjensidigestiftelsen (Unknown); Stiftelsen Helse og Rehabilitering (Other); Organisasjonen Voksne for Barn (Unknown)
Responsible Party: Principal Investigator, Samira Lekhal, MD, PhD, Head Children department Morbid Obesity Center, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FamilY
Record Dates: First submitted 2010-04-21; First posted 2010-04-26 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Obesity; Child; Parent; Family
MeSH Terms: conditions — Obesity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - family camp (Experimental): Obese families participate in a two week camp with two years follow-up.
  Interventions: Behavioral: Parent Management Training - Oregon (PMTO); Behavioral: Motivational interviewing; Behavioral: Dynamic group therapy
- Group B - family lifestyle school (Other): Families participate in a four day practical course about lifestyle.
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Parent Management Training - Oregon (PMTO) — Method to help parents and caregivers manage the behavior of the children they are responsible for.
  Arms: Group A - family camp
Behavioral: Motivational interviewing — Communication method to facilitate behavioral change and empower the parents.
Behavioral: Dynamic group therapy — Focuses on individual experiences within families and/or parents/children, and that the participants are their own experts.
  Arms: Group A - family camp

SUMMARY:
The study compares the effect on BMI of two different treatment options for obesity in childhood. Families with at least one obese child and parent are invited to join the project. The hypothesis is that family camp gives an additional reduction in BMI compared to a less intensive family lifestyle school.

DETAILED DESCRIPTION:
Participants are randomised to two intervention groups:

A): Two weeks family camp and two years follow-up as a cooperation with primary health care, private rehabilitation center and specialist health care.

B): Four days lifestyle school with two years follow-up as a cooperation with primary health care and specialist health care

ELIGIBILITY:
Inclusion Criteria:

* age 7 to 12 years
* BMI > iso-BMI 30 (Coles index)

Exclusion Criteria:

* syndromatic obesity
* obesity related to diseases
* local community not involved
* child has present follow-up because of obesity in secondary health care
* parent has present/planned follow-up because of obesity in secondary health care

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2013-05 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
BMI-SDS | After 2 years
  Primary Outcome Measure is body mass index-standard deviation score. Reduced values from baseline to endpoint means reduced overweight.

SECONDARY OUTCOMES:
Quality of life | After 2 years
  Questionnaire for children and parent
Physical fitness | After 2 years
  Six minutes walk test for children and parents.
Behaviour | After 2 years
  Evaluating effect of intervention on risk for psyciatric disorders.
Blood samples | After 2 years
  Improvement in spesific blood tests with relevance to metabolic syndrome after 2 years intervention? Blood is biobanked at baseline and after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Lekhal, PhD, MD, Principal Investigator — The Hospital of Vestfold; Jøran Hjelmesæth, PhD, MD, Study Chair — The Hospital of Vestfold
Locations (2):
- Norway (2):
  - St Olavs Hospital, Trondheim
  - Morbid Obesity Center, The Hospital of Vestfold, South-Eastern Norway Regional Health Authority, Tønsberg

REFERENCES:
- [Derived] Benestad B, Karlsen TI, Smastuen MC, Lekhal S, Hertel JK, Steinsbekk S, Kolotkin RL, Odegard RA, Hjelmesaeth J. Health-related quality of life after camp-based family obesity treatment: an RCT. BMJ Paediatr Open. 2019 Apr 3;3(1):e000413. doi: 10.1136/bmjpo-2018-000413. eCollection 2019. PMID 31206074
- [Derived] Benestad B, Lekhal S, Smastuen MC, Hertel JK, Halsteinli V, Odegard RA, Hjelmesaeth J. Camp-based family treatment of childhood obesity: randomised controlled trial. Arch Dis Child. 2017 Apr;102(4):303-310. doi: 10.1136/archdischild-2015-309813. Epub 2016 Nov 2. PMID 27806969